CLINICAL TRIAL: NCT02702284
Title: Advance Directives Completion Rates and an Intervention to Address Health Literacy in a Clinic Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB201500776
Record Dates: First submitted 2016-02-29; First posted 2016-03-08 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Health Literacy
Keywords: Advance Directives; Healthcare power of attorney
MeSH Terms: interventions — Advance Directives; Living Wills; Insemination, Artificial, Heterologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Adequate health literacy, control (Other): This group of subjects will be referred to clinic staff for assistance with the advance directives (AD) and will not receive assistance from a research assistant. In addition, the research assistance will ask questions regarding the information received for the AD.
  Interventions: Behavioral: Advance Directives without assistance
- Adequate health literacy, intervention (Experimental): The subjects in this group will hear a research assistant review the advance directive and be offered an opportunity to watch a video about advance directives.
  Interventions: Behavioral: Advance Directives
- Limited health literacy, control (Other): This group of subjects will be referred to clinic staff for assistance with the advance directives (AD) and will not receive assistance from a research assistant. In addition, the research assistance will ask questions regarding the information received for the AD.
  Interventions: Behavioral: Advance Directives without assistance
- Limited health literacy, intervention (Experimental): The subjects in this group will hear a research assistant review the advance directive and be offered an opportunity to watch a video about advance directives.
  Interventions: Behavioral: Advance Directives

INTERVENTIONS:
Behavioral: Advance Directives — These subject's will have a research assistant (RA) review and walk through the advance directives brochure. The RA will read all of the brochure to the patient and prompt for questions. In addition, a link to an educational video on advance directives. The advance directive link will be either texted or emailed or given in paper per the subject's preference.
  Other Names: Living will
  Arms: Adequate health literacy, intervention; Limited health literacy, intervention
Behavioral: Advance Directives without assistance — This group of subjects will be provided with the advance directive and then referred to clinic staff for assistance.
  Other Names: Living will
  Arms: Adequate health literacy, control; Limited health literacy, control

SUMMARY:
The ability to communicate with patients is profoundly impacted by their health literacy - the ability to interpret documents, read and write prose, use quantitative information and speak and listen effectively. Limited health literacy is commonplace and associated with multiple poor health outcomes including frequent readmission's and high mortality. Advance directives are an important tool in respecting patient autonomy in health care interventions. Advance directives can also reduce health care costs by avoiding unwanted, unnecessary care at the end of life. At the University of Florida (UF) Health currently an initiative is underway to improve the delivery of advance directives to patients in the hospital as well as the outpatient clinics.

The aim of this research study is to enhance completion rates of advance directives by taking into consideration a patient's health literacy level. Specifically, the investigators plan to assess the impact of an ambulatory intervention on the completion rate of advance directives for patients with adequate and limited health literacy. The hypothesis is that both groups (adequate and limited health literacy) will benefit from the intervention, but patients with limited health literacy will show a greater improvement in the advance directives completion rate.

DETAILED DESCRIPTION:
The purpose of this research study is to improve completion of Advance Directives. These are documents that patients use to let doctors know what their wishes for treatment are and who they would want to make decisions for them if they could not make decisions for themselves.

At the time of the clinic visit to the Internal Medicine at Medical Plaza (IMMP) or the Internal Medicine at Tower Hill (IMTH) subjects will be invited to participate in the study.

Research Assistant(s) RA Responsibilities:

All Potential Study Subjects:

1. RA will interview study subject in a private area (exam room or empty office).
2. RA will assess eligibility criteria.
3. RA will obtain informed consent.
4. RA will randomize the subjects to either intervention or control.
5. RA will explain to the subjects how to return the advance directive (AD)

For the Intervention group:

1. RA will review and walk through the University of Florida (UF) AD brochure
2. RA will offer subjects a link to a patient education video on advance directives. The link will be texted or emailed or given in paper per the subject's preference.
3. RA will conduct a brief satisfaction questionnaire addressing the activity review of the UF AD brochure.
4. RA will ask

   1. Did addressing advance directives enhance today's experience at the clinic?
   2. Do you think that advance directives be routinely addressed at visits to the doctor?

Control group:

If the subject is ready to complete an advance directive they will be referred to clinic staff for assistance.

RA will ask

1. Did addressing advance directives enhance today's experience at the clinic?
2. Do you think that advance directives should be routinely addressed at visits to the doctor?

ELIGIBILITY:
Inclusion Criteria:

* No advance directive in electronic medical record,
* speaks English,
* has intact cognitive function

Exclusion Criteria:

* Age 50 or under,
* already has an advance directive in electronic medical record,
* does not speak English,
* cognitive dysfunction

Min Age: 51 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Presence of advance directive scanned into electronic medical record | 6 months from enrollment
  The research assistant will review the subject's electronic medical record for a copy of a signed advance directive.

SECONDARY OUTCOMES:
Number of reminder phone calls needed | 6 months
  1. All subjects' charts will be reviewed to see if the subjects have submitted AD.
  2. If a subject has not submitted an AD, the RA will remind them to return their advance directive papers via phone call 1, 3 and 5 months after they are enrolled
Client Evaluation of Services Questionnaire | day of study
  Score 8 - 32
  1. How would you rate the quality of services you have received at your visit today?
  2. Did you get the kind of service you wanted?
  3. To what extent has your visit met your needs?
  4. If a friend were in need of similar help, would you recommend our office to him or her?
  5. How satisfied are you with the amount of help you have received?
  6. Have the services you receive helped you to deal more effectively with your problems?
  7. In an overall, general sense, how satisfied are you with the service you have received at the visit?
  8. If you were to seek help again, would you come back to our office?
  9. Did addressing Advance Directives enhance your clinic experience today?
  10. Do you think Advance Directives should be routinely addressed at your doctor's visit?

CONTACTS AND LOCATIONS:
Overall Officials: Melanie G Hagen, MD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Tower Hill Internal Medicine, Gainesville, Florida
  - Internal Medicine at Medical Plaza, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barker PC, Holland NP, Shore O, Cook RL, Zhang Y, Warring CD, Hagen MG. The Effect of Health Literacy on a Brief Intervention to Improve Advance Directive Completion: A Randomized Controlled Study. J Prim Care Community Health. 2021 Jan-Dec;12:21501327211000221. doi: 10.1177/21501327211000221. PMID 33719708